CLINICAL TRIAL: NCT01911624
Title: Direct Thrombin Inhibitors Versus LMWH in Staphylococcus Aureus Bacteraemia. A Prospective Randomized Controlled Academic Single-centre Feasibility Study.
Brief Title: Direct Thrombin Inhibitors Versus LMWH in Staphylococcus Aureus Bacteraemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Peter Verhamme, Prof., Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: S54881
Record Dates: First submitted 2013-06-14; First posted 2013-07-30 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Staphylococcus Aureus Bacteraemia
MeSH Terms: interventions — Dabigatran; argatroban; Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- direct thrombin inhibition (Experimental): dabigatran 110 mg BID, po argatroban (0.5 - 1 µg/kg/min) if peroral therapy is not possible
  Interventions: Drug: direct thrombin inhibition
- enoxaparin (Active Comparator): enoxaparin 40 mg od, sc
  Interventions: Drug: enoxaparin

INTERVENTIONS:
Drug: direct thrombin inhibition
  Other Names: dabigatran; argatroban
  Arms: direct thrombin inhibition
Drug: enoxaparin
  Other Names: clexane
  Arms: enoxaparin

SUMMARY:
Safety and efficacy of direct thrombin inhibitors versus enoxaparin in patients with staphylococcus aureus bacteraemia.

The study hypothesizes that inhibition of the coagulase-activity of S. aureus by direct thrombin inhibitors is safe and translates into a better outcome of patients with S. aureus bacteremia.

DETAILED DESCRIPTION:
Single center randomized controlled trial of direct thrombin inhibitors versus standard enoxaparin.

* Feasibility: proportion of patients eligible for randomization; clinically attained concentration of DTI and resulting staphylothrombin inhibition
* Safety: bleeding events (major/ clinically relevant non-major)
* Efficacy: thrombotic events during the thromboprophylactic treatment + 3 days
* Secondary outcome measures

  * Coagulation parameters: evolution of D-dimers from day 0-4; other lab parameters of coagulation (PT/APTT/fibrinogen/platelet count)
  * Inflammatory parameters: CRP, white blood cell count, neutrophilia
  * Clinical outcomes: metastatic infections, assessed clinically or by PET/CT; relapse of S. aureus bacteremia; defervescence; persistent positive blood cultures; hospital stay, mortality.

ELIGIBILITY:
Inclusion Criteria:

* Positive blood culture for staphylococcus aureus
* Symptoms or signs of infection
* Indication for thromboprophylaxis

Exclusion Criteria:

* Contraindication for thromboprophylaxis
* Significant active bleeding or risk of excessive bleeding
* Heparin-induced thrombocytopenia
* Severe liver and kidney disease
* Pregnancy and lactation.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2013-01; Primary Completion 2016-04 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Primary Safety Outcome is the occurence of clinically-relevant bleeding events | From date of randomization up to end of study drug + 3 days

SECONDARY OUTCOMES:
The primary efficacy outcome is the occurence of metastatic infection | From randomization until month 3
  as documented with a PET-CTscan in eligible patients on D7-10 or clinically-overt metastatic infectious foci

OTHER OUTCOMES:
Laboratory markers of coagulation | From randomization until D7-10
  D-dimeren, fibrinogen, APTT, PT dabigatran level or antiXa
Laboratory markers of inflammation | From randomization until D7-10
  CRP
Clinical outcomes after S. aureus bacteremia | From randomization until M3

CONTACTS AND LOCATIONS:
Overall Officials: Peter Verhamme, Doctor, Principal Investigator — Bloedings-en vaatziekten, UZ Gasthuisberg
Locations (1):
- KUleuven/UZ Gasthuisberg, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided